CLINICAL TRIAL: NCT05022966
Title: The Relationship Between Physical Activity and Falling Risk and Fear of Falling in Elderlies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Assist. Prof., Izmir Bakircay University
Other Study IDs: 2021-06-277
Record Dates: First submitted 2021-08-22; First posted 2021-08-26 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Healthy Aging
Keywords: Physical activity; Daily life activities; Fear of falling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older people
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Individuals did not received any intervention.

SUMMARY:
Aging is a physiological process, and it is a picture in which a decrease in physical functions, regression in cognitive abilities, decrease in social activities, loss of functionality in their lives occur and these are accompanied by many health problems. As a result of the changes in the human body and mind, the productivity of the organism and the ability of the person to adapt to the environment decrease. According to the data of the World Health Organization, this period is considered to be 65 years and over, and according to the data of the United Nations, 60 years and over.

The aim of this study is to investigate the effect of physical activity level on activities of daily living and fear of falling in elderlies.

DETAILED DESCRIPTION:
Physical activity is defined as voluntary movements produced by skeletal muscles that result in increased energy expenditure. Physical activity includes activities that are done as a part of daily life. One of the protective factors against mental and physical diseases in old age is physical activity. There is a linear and strong link between physical activity and health. Physical inactivity accounts for 6% of deaths worldwide and ranks fourth among risk factors. Being physically active has an important place in the protection and development of health, active healthy aging, and protection from diseases caused by inactivity.

Activities of daily living are essential and important vital functions for a healthy or sick individual to survive. The most important wishes of aging individuals are to be able to perform daily living activities such as walking, climbing stairs, and getting up without the need for help. The activities of daily living of the elderly are reduced or prevented, and they begin to lose their independence.

Fear of falling, which is frequently encountered in the elderly, is among the psychological consequences of falling. Fear of falling, which is defined as avoidance of activity or fear of falling leading to decreased activity, is seen in 35-55% of the elderly. Falls are among the most common causes of morbidity and mortality in the elderly. One-third of people over the age of 65 fall each year, and half of the falls are recurrent falls. Depending on the fear of falling, the physical activities of the elderly may be restricted.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being 60 years old or older
* Staying in a nursing home for at least 1 month
* Independent mobilization of the participants

Exclusion Criteria:

* Having a problem that prevents communication
* Having multiple comorbidities
* Having a cognitive problem

Ages: 60 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study group of this research is planned to be composed of residents of Melmira Elderly Care Center and Nursing Home.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Scale For Elderly | At baseline
  Physical Activity Scale For Elderly (PASE) includes participants' walking, mild, moderate, vigorous sports and recreational activities, muscle strength and endurance exercises, work-related activities including walking and standing, lawn and garden maintenance, caring for another person, home repairs, heavy-duty sports and recreational activities in the past week. Home and work-related activities are scored as yes or no. For work-related activities, paid or unpaid work is scored in hours per week. The total PASE score is calculated by multiplying the time spent in each activity (hours per week) or participation in an activity (ie yes or no) by the experimentally derived item weights, and then adding the overall activities. The overall PASE score ranges from 0 to 400 or more, with higher scores indicating better levels of physical activity.
Modified Barthel Index | At baseline
  Modified Barthel Index is a 10-item scale that evaluates physical independence in activities of daily living (transfer, ambulation/wheelchair use, stair climbing, feeding, dressing, self-regulation, bathing, toilet use, urinary continence, stool continence). The total score (0-100) is calculated by scoring each item separately with a three-digit scoring system. The total score ranges from 0 to 100, where "0" indicates complete dependency and "100" indicates complete independence. The sensitivity of the index was increased by using a five-step scoring system in the Modified Barthel index modified by Shah.
Falls Efficacy Scale International | At baseline
  Fall Effectiveness Scale-International (FES-I), developed and approved by the European Fall Prevention Network (ProFaNE), has become a widely accepted tool for assessing fall anxiety. The FES-I is a self-reported questionnaire that provides information on the level of anxiety about falls for a range of activities of daily living. The original questionnaire contains 16 items scored on a four-point scale (1 = not at all interested to 4 = very interested). The lowest score that can be obtained from the survey is 16 and the highest score is 64. A high score indicates an increased level of anxiety. The Turkish validity and reliability of the questionnaire was performed by Ulus et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No